CLINICAL TRIAL: NCT00239070
Title: A Prospective, Open-label, Multicenter, International Follow-up Study on the Safety and Efficacy of Enteric-coated Mycophenolate Sodium (EC-MPS) in Kidney Transplant Recipients
Brief Title: Extension Study on the Safety and Efficacy of Enteric-coated Mycophenolate Sodium in Kidney Transplant Recipients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Novartis, Novartis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CERL080A2405IN01E1
Record Dates: First submitted 2005-10-12; First posted 2005-10-14 (Estimated); Last update posted 2011-01-31 (Estimated); Status verified 2011-01

CONDITIONS: Renal Transplantation
Keywords: EC-MPS, renal transplantation, de novo patients

INTERVENTIONS:
Drug: Enteric-Coated Mycophenolate Sodium (EC-MPS)

SUMMARY:
This extension study is to assess the long-term safety of EC-MPS

ELIGIBILITY:
Inclusion / Exclusion Criteria - All patients who completed study CERL080A2405-IN01 and who are willing to continue treatment with Enteric-Coated Mycophenolate Sodium.

Other protocol-defined inclusion / exclusion criteria may apply

-

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2003-04; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
To assess patient and graft survival, acute rejection incidence, graft function and specific pertinent safety parameters in de novo renal transplant recipients.

SECONDARY OUTCOMES:
To assess the respective influence of parameters (demographic characteristics, transplant-related variables, medical conditions and post-transplantation complications) on clinical outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis